CLINICAL TRIAL: NCT07012421
Title: Comparison of Community and Hospital Antibiotic Use Practices, Susceptibility and ResisTance and Determinants of Care Seeking Among Patients With Urinary Tract Infections (CAST-UTI)
Brief Title: Community Antibiotic Use, Susceptibility and ResisTance Among Patients With Urinary Tract Infections (CAST-UTI)
Acronym: CAST-UTI
Status: Recruiting | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: Makerere University (Other); Infectious Diseases Research Collaboration, Uganda (Other)
Responsible Party: Sponsor
Other Study IDs: 2024.0149; 226461/Z/22/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2024-12-22; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-12

CONDITIONS: Urinary Tract Infections (UTIs)
Keywords: Low- and middle-income countries; Uganda; antibiotic resistance; urinary tract infection; multidrug resistant organisms
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine sample and perianal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Namuwongo community: The Namuwongo informal settlement is located in the urban area of Kampala, Uganda. An estimated 70% of residents in the informal settlement routinely (within the last month) use antibiotics. Houses are overcrowded with residents paying to use public toilets.
  The investigators are recruiting from community drug retail outlets and the outpatient department of Kitsugu health centre located next to Namuwongo.
- Muyenga community: The Muyenga and Bukasa neighbourhoods are also located in the urban area of Kampala, Uganda, but is more affluent than the Namuwongo informal settlement. Residents in Muyenga can afford more expensive treatments at community drug retail outlets (CDROs)/clinics.
  The investigators are recruiting from community drug retail outlets and the outpatient department of Naguru hospital located next to Muyenga and Bukasa neighbourhoods.

SUMMARY:
1. General objective

   This pilot study aims to compare the prevalence of resistance in bacteria causing UTIs among patients seeking care outside the hospital settings (CDROs) to the WHO-GLASS data.
2. Specific objectives

2-1 Primary objectives:

* Determine the resistance profiles of uropathogens and carriage strains from patients with uncomplicated UTIs attending community drug retail outlets (CDRO's) and in hospitals*.
* Compare the resistance profiles of the uropathogens from patients with uncomplicated UTIs attending CDROs and hospitals to those in the WHO-GLASS database.
* Explore the patient pathway and its impact on antibiotic use among patients presenting to CDROs and hospitals with uncomplicated UTIs.
* Determine the appropriateness of antimicrobial use in the treatment of uncomplicated UTIs among patients presenting to CDROs and hospitals

2-2 Secondary objectives:

* Compare resistance profiles among the uropathogens from patients from two neighbourhoods in Kampala.
* Examine environmental samples between the study sites to determine the presence of antibiotic residues and AMR two neighbourhoods in Kampala.

ELIGIBILITY:
Inclusion criteria:

* Must have one or more of the following clinical presentations regardless of age:

acute (< 2 weeks) dysuria. increased urinary urgency and frequency, irritation, discharge. increased lower abdominal pain or discomfort and sometimes gross haematuria.

* In elderly patients with pre-existing urinary symptoms: increased acute urinary changes.

Exclusion criteria:

* People without symptoms of UTI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting with acute UTIs arriving in CDROs/clinics and hospitals within the boundaries of the two study communities are eligible to enrol (Namuwongo informal settlement, Muyenga, and Bukasa neighbourhoods) during the 12-month study collection period.
  Workers from CDROs and healthcare clinics/ hospital outpatient departments from the same two communities will be asked to complete the surveys.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-10-06 (Actual); Primary Completion 2025-10-05 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
A comparison of resistance profiles between GLASS and community uropathogens in Uganda | At the end of 12 months data collection
  Twelve-month prevalence of antimicrobial resistance in Escherichia coli and Klebsiella pneumoniae isolates causing urinary tract infections, comparing GLASS surveillance data and data collected in the community in Uganda. Resistance will be measured as the proportion of isolates non-susceptible to key antibiotic classes (e.g., third-generation cephalosporins, fluoroquinolones, carbapenems).

SECONDARY OUTCOMES:
Patient pathway and antibiotic use in the community | 28 days
  Characterisation of the patient pathway from symptom onset to days 7 and 28 in individuals with urinary tract infections, and its association with antibiotic use patterns (e.g., timing, type, source, appropriateness).
  Collect information on healthcare seeking behaviour for eligible patients, including their sociodemographic information, antibiotics purchased, and cost of antibiotics.
Appropriateness of antimicrobial use in the treatment | 7 days after enrolment
  Proportion of UTI cases in the community with microbiologically confirmed E. coli or K. pneumoniae where the prescribed or obtained antibiotic treatment was appropriate, based on standard treatment guidelines and the organism's resistance profile.
Retail outlet determinants of treating healthcare-seeking among patients with suspected UTIs | At the end of 12 months after enrolment
  The investigators are collecting information on the number of UTIs presenting at community drug retail outlets over twelve months, antibiotic availability in the ommunity drug retail outlet, compliance with regulations, and healthcare worker training level.
Antibiotic residues and AMR in two neighbourhoods in Kampala | Once a month for 12 months after study commencement
  Detection of antibiotic residues and antimicrobial resistant organisms in environmental water samples from channels linking the two study neighbourhoods.
  Through detection of antibiotic residues and testing of microorganisms isolated from the waterway and sediment.

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Diseases Research Collaboration (IDRC), Uganda, Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: No
IPD would contain identifiable personal information. Therefore, the anonymised data will be collected through REDCap which is a secure data management tool.

REFERENCES:
- [Background] Gebremariam G, Legese H, Woldu Y, Araya T, Hagos K, GebreyesusWasihun A. Bacteriological profile, risk factors and antimicrobial susceptibility patterns of symptomatic urinary tract infection among students of Mekelle University, northern Ethiopia. BMC Infect Dis. 2019 Nov 8;19(1):950. doi: 10.1186/s12879-019-4610-2. PMID 31703645
- [Background] Flores-Mireles AL, Walker JN, Caparon M, Hultgren SJ. Urinary tract infections: epidemiology, mechanisms of infection and treatment options. Nat Rev Microbiol. 2015 May;13(5):269-84. doi: 10.1038/nrmicro3432. Epub 2015 Apr 8. PMID 25853778
- [Background] Cambaco O, Alonso Menendez Y, Kinsman J, Sigauque B, Wertheim H, Do N, Gyapong M, John-Langba J, Sevene E, Munguambe K. Community knowledge and practices regarding antibiotic use in rural Mozambique: where is the starting point for prevention of antibiotic resistance? BMC Public Health. 2020 Jul 29;20(1):1183. doi: 10.1186/s12889-020-09243-x. PMID 32727445
- [Background] Mbonye AK, Buregyeya E, Rutebemberwa E, Clarke SE, Lal S, Hansen KS, Magnussen P, LaRussa P. Prescription for antibiotics at drug shops and strategies to improve quality of care and patient safety: a cross-sectional survey in the private sector in Uganda. BMJ Open. 2016 Mar 15;6(3):e010632. doi: 10.1136/bmjopen-2015-010632. PMID 26980439
- [Background] Frost I, Kapoor G, Craig J, Liu D, Laxminarayan R. Status, challenges and gaps in antimicrobial resistance surveillance around the world. J Glob Antimicrob Resist. 2021 Jun;25:222-226. doi: 10.1016/j.jgar.2021.03.016. Epub 2021 Apr 15. No abstract available. PMID 33845163
- [Background] Collignon PJ, McEwen SA. One Health-Its Importance in Helping to Better Control Antimicrobial Resistance. Trop Med Infect Dis. 2019 Jan 29;4(1):22. doi: 10.3390/tropicalmed4010022. PMID 30700019
- [Background] Collignon P, Beggs JJ. Socioeconomic Enablers for Contagion: Factors Impelling the Antimicrobial Resistance Epidemic. Antibiotics (Basel). 2019 Jun 30;8(3):86. doi: 10.3390/antibiotics8030086. PMID 31261988
- [Background] Antimicrobial Resistance Collaborators. Global burden of bacterial antimicrobial resistance in 2019: a systematic analysis. Lancet. 2022 Feb 12;399(10325):629-655. doi: 10.1016/S0140-6736(21)02724-0. Epub 2022 Jan 19. PMID 35065702